CLINICAL TRIAL: NCT00254735
Title: Quetiapine Augmentation in Severe Obsessive Compulsive Disorder (OCD) - Pilot Study
Brief Title: Quetiapine Augmentation in Severe Obsessive Compulsive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5077/9059; D1441C09059
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive Compulsive Disorder (OCD)
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: quetiapine fumarate
Drug: SSRI/Clomipramine

SUMMARY:
The purpose of the study is to evaluate the efficacy of quetiapine or placebo added to baseline treatment of SSRI/clomipramine for the treatment of OCD in adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, men and women aged ³18 to £65 years with diagnosis of OCD, at least 12 weeks of treatment with SSRI or clomipramine

Exclusion Criteria:

* Substance abuse or dependence, female patients who are pregnant, lactating or at risk of pregnancy, known intolerance or lack of response to quetiapine, use of antihypertensive medication with changing doses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2002-04; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Absolute change of OCD symptoms from baseline to endpoint on the total Y-BOCS score.

SECONDARY OUTCOMES:
Change of comorbid psychiatric symptoms and measures of quality of life from baseline to endpoint documented by different scales.
Evaluation of the safety and tolerability profile of quetiapine compared to placebo added to a baseline medication of SSRI/clomipramine.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Germany Medical Director, MD, Study Director — AstraZeneca
Locations (2):
- Germany (2):
  - Research Site, Freiburg im Breisgau
  - Research Site, Lübeck